CLINICAL TRIAL: NCT00488280
Title: Restoring Walking in Non-ambulatory Children With Severe Chronic SCI (Kids STEP Study)
Brief Title: Restoring Walking in Non-ambulatory Children With Severe Chronic Spinal Cord Injury (SCI) (Kids STEP Study)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Brooks Rehabilitation (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 313-2006
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: walking; walking recovery; physical therapy; locomotor training; body weight support; neuroplasticity; step; treadmill; treadmill training; locomotion
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kids Step Study: Locomotor Training: All children who participate will be in the experimental cohort, KSS-#, and receive 60 sessions of daily locomotor training. This experimental cohort will also undergo clinical and neurophysiological testing pre, during, and post 60 sessions of locomotor training.
  Interventions: Behavioral: Locomotor Training

INTERVENTIONS:
Behavioral: Locomotor Training — Task-specific practice of walking with assistance from trainers using body weight support and treadmill followed by training over ground, 5x/week, approximately 1.5 hours/day
  Other Names: body weight supported treadmill training; activity-based therapy

SUMMARY:
The Kids STEP Study aims to

1. Determine if walking can be restored in children with incomplete SCI and little to no leg movement
2. Identify the neural pathways that permit recovery of walking

DETAILED DESCRIPTION:
Locomotor training (LT) is an activity-based therapy to promote plasticity and recovery of walking. It is based on animal studies investigating walking recovery after spinal cord injury and the nervous system's control of walking. Normal walking is achieved through the interaction of multiple levels of the neural axis (cortex, brain stem, spinal cord). However, a basic rhythmic walking pattern is generated by central pattern generators (CPGs) located within the spinal cord. Investigations of central pattern generators indicate that sensory input specific to the task of walking can enhance the firing of these spinal neuronal centers. Thus, LT is an intensive walking program designed to provide sensory input to the spinal cord so that the neural output from the spinal CPGs can be maximized. In addition, LT uses a treadmill and a harness to provide partial body weight support enabling persons with injury to repetitively practice walking in a safe, enabling environment.

Children enrolled in the study (after medical clearance and consent to participate) will undergo extensive testing and complete 12 weeks of locomotor training. Testing will examine the child's neurologic and functional status. Tests to examine functional status include: ASIA evaluation of sensory and motor function, gait analysis, comprehensive strength tests, and assessment of skills such as cycling, stepping, and kicking. Tests to examine the child's neurologic injury include: MRI, Transcranial Magnetic Stimulation (TMS), and reflex testing. Locomotor training will be conducted daily (5 days/ week) for a total of 60 sessions over 12 weeks. During training children will work closely with therapists, researcher, and trainers to practice walking skills on the treadmill and over-ground.

ELIGIBILITY:
Inclusion Criteria:

Individuals with SCI will include:

* Pre-adolescent children, ages 3-13 yrs old
* A diagnosis of first time, non-progressive SCI, upper motor neuron lesion, including, but not limited to, etiology from trauma, inflammation, vascular, surgical re-section due to localized tumor removal or orthopedic pathology resulting in clinical signs of lower cervical or thoracic spinal cord injury
* Non-ambulatory or impaired ambulation for greater than 1 yr, such that physical assistance and the use of assistive devices (i.e. walker) and/or leg braces (i.e. knee- ankle- foot orthoses (KAFOs)) are required to ambulate
* A SCI as defined by the American Spinal Injury Association (ASIA) Impairment Scale category B or C
* A medically stable condition that is asymptomatic for bladder infection, decubiti, osteoporosis, cardiopulmonary disease, pain, or other significant medical complications that would prohibit or interfere with testing of walking function and training or alter compliance with a training protocol
* Documented medical approval from the participant's personal physician verifying the participant's medical status
* Parent's informed consent for children

Exclusion Criteria

Children with SCI who -

* Are currently participating in a rehabilitation program or another research protocol that could interfere or influence the outcome measures of the current study
* Have a history of congenital SCI (e.g. Chiari malformation, myelomeningocele, intraspinal neoplasm, Frederich's ataxia) or other degenerative spinal disorders (e.g. spinocerebellar degeneration or syringomyelia) that may complicate the treatment and/or evaluation procedures
* Children who are diabetic or have implants, pacemakers, or devices which are not NMR/MRI compatible and are not suitable for the study

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with SCI for whom walking recovery is unlikely
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Recovery of walking, assessed in treadmill/ BWS environment and overground | pre-training, after 20, 40, and 60 sessions of locomotor training

SECONDARY OUTCOMES:
Amount of daily step activity | during and post 60 sessions of locomotor training
Walking independence, WISCI II | during and post 60 sessions of locomotor training
Stepping assessment and kinematic analysis | Post 20, 40, and 60 sessions of locomotor training
Analysis of locomotor tasks such as crawling, swimming, cycling | post 20, 40, and 60 sessions of locomotor training
Self-selected and fast gait speed | Pre-training and after 20, 40, 60 sessions (post-LT)
Spinal MRI to assess injury | Pre-training
Spinal reflex assessment (H reflex) | Pre-training and post-training
Correlation of locomotion recovery and isolated voluntary leg movement (ASIA motor score) | Pre-training and post-training
Correlation and assessment of reticulospinal tract (Acoustic startle reflex)with recovery of locomotion | Pre-training and post-training
Correlation and assessment of corticospinal tract integrity via transcranial magnetic stimulation | Pre-training and post-training

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Behrman, PhD, PT, Principal Investigator — University of Florida; Dena R Howland, PhD, OT, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Barbeau H, Nadeau S, Garneau C. Physical determinants, emerging concepts, and training approaches in gait of individuals with spinal cord injury. J Neurotrauma. 2006 Mar-Apr;23(3-4):571-85. doi: 10.1089/neu.2006.23.571. PMID 16629638
- [Background] Barbeau H, Ladouceur M, Norman KE, Pepin A, Leroux A. Walking after spinal cord injury: evaluation, treatment, and functional recovery. Arch Phys Med Rehabil. 1999 Feb;80(2):225-35. doi: 10.1016/s0003-9993(99)90126-0. PMID 10025502
- [Background] Behrman AL, Lawless-Dixon AR, Davis SB, Bowden MG, Nair P, Phadke C, Hannold EM, Plummer P, Harkema SJ. Locomotor training progression and outcomes after incomplete spinal cord injury. Phys Ther. 2005 Dec;85(12):1356-71. PMID 16305274
- [Background] Behrman AL, Harkema SJ. Locomotor training after human spinal cord injury: a series of case studies. Phys Ther. 2000 Jul;80(7):688-700. PMID 10869131
- [Background] Edgerton VR, Tillakaratne NJ, Bigbee AJ, de Leon RD, Roy RR. Plasticity of the spinal neural circuitry after injury. Annu Rev Neurosci. 2004;27:145-67. doi: 10.1146/annurev.neuro.27.070203.144308. PMID 15217329
- [Background] Behrman AL, Bowden MG, Nair PM. Neuroplasticity after spinal cord injury and training: an emerging paradigm shift in rehabilitation and walking recovery. Phys Ther. 2006 Oct;86(10):1406-25. doi: 10.2522/ptj.20050212. PMID 17012645
- [Derived] Howland DR, Trimble SA, Fox EJ, Tester NJ, Spiess MR, Senesac CR, Kleim JA, Spierre LZ, Rose DK, Johns JS, Ugiliweneza B, Reier PJ, Behrman AL. Recovery of walking in nonambulatory children with chronic spinal cord injuries: Case series. J Neurosci Res. 2023 Jun;101(6):826-842. doi: 10.1002/jnr.25162. Epub 2023 Jan 23. PMID 36690607